CLINICAL TRIAL: NCT06393192
Title: Postoperative Analgesic Effects of Various Quadratus Lumborum Block Approaches Following Cesarean Section.
Brief Title: The Post Cesarean Section Analgesic Effect of Various Quadratus Lumborum Block Approaches
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hatem Awaga, Lecturer of Obstetrics and Gynecology, Sohag University
Other Study IDs: Soh-Med-23-09-6PD
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Painless Labor; Epidural Analgesia; Cesarean Section
MeSH Terms: interventions — Analgesia, Epidural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Epidural analgesia (EA) only group: In this group 20 patients fulfilling the eligibility criteria, the epidural needle was inserted at the level of the intervertebral gap that separates the 2nd & 3rd spinal bones.
  Upon locating the epidural space through the utilization of the loss of resistance to saline approach, the tip of a spinal needle was inserted through the epidural needle. In order to reach a specific level of sensory block up to the sixth thoracic dermatome, each pregnant woman was administered intrathecal anesthetic consisting of 0.75 percent bupivacaine in a volume of 1.3-1.7 milliliter.
  Subsequently, we removed the needle & proceeded to place an epidural catheter through the epidural needle as a precautionary measure in the event of intrathecal anesthetic failure. The EA group received a single dosage of six milliliters of saline solution containing nine milligrams of bupivacaine (0.15%) & 2 mg of morphine via the epidural catheter for postoperative pain management.
  Interventions: Procedure: Epidural analgesia (EA) only group
- Quadratus Lumborum 2 (QL2) group: In this group 20 patients fulfilling the eligibility criteria, the ultrasound transducer was positioned horizontally at the level of L2-3 on both sides of the body. It was adjusted until the "Shamrock sign" created by the QL muscle, psoas major, and erector spinae was visible. The imaging depth was set among 0 as well as 9.9 cm. Needles were inserted from the front-lateral to back-medial direction. An injection of local anesthetic was administered behind the QL muscle.0.2% bupivacaine were administered at a volume of thirty milliliters at the specified sites on each side, resulting in a total of Sixty mL
  Interventions: Procedure: Quadratus lumborum block (QL2)
- Quadratus Lumborum 3 (QL3) group: In this group 20 patients fulfilling the eligibility criteria, the ultrasound transducer was positioned horizontally at the level of L2-3 on both sides of the body. It was adjusted until the "Shamrock sign" created by the QL muscle, psoas major, and erector spinae was visible. The imaging depth was set among 0 as well as 9.9 cm. Needles were inserted from the front-lateral to back-medial direction. An injection of local anesthetic was administered among the QL and the psoas major muscles.0.2% bupivacaine were administered at a volume of thirty milliliters at the specified sites on each side, resulting in a total of Sixty mL
  Interventions: Procedure: Quadratus lumborum block 3(QL3)
- Quadratus Lumborum 2+3 (QL2+3) group: In this group 20 patients fulfilling the eligibility criteria, the QL2+3 block can be performed in a single plane with only one puncture on each side. 0.2 percent bupivacaine solution of fifteen milliliters were administered at each injection site, with the needle being inserted once on each side
  Interventions: Procedure: Quadratus lumborum block 2+3 QL(2+3)

INTERVENTIONS:
Procedure: Epidural analgesia (EA) only group — The epidural needle will be inserted into the lumbar epidural space at the level of L2-3 intervertebral space.
  Groups: Epidural analgesia (EA) only group
Procedure: Quadratus lumborum block (QL2) — 0.2% bupivacaine at a volume of thirty milliliters were administered at the specified sites on each side behind the QL muscle, resulting in a total of Sixty mL
  Groups: Quadratus Lumborum 2 (QL2) group
Procedure: Quadratus lumborum block 3(QL3) — 0.2% bupivacaine at a volume of thirty milliliters were administered at the specified sites on each side among the QL muscle and the psoas major, resulting in a total of Sixty mL
  Groups: Quadratus Lumborum 3 (QL3) group
Procedure: Quadratus lumborum block 2+3 QL(2+3) — 0.2 percent bupivacaine solution of fifteen milliliters were administered at each injection site, with the needle being inserted once on each side
  Groups: Quadratus Lumborum 2+3 (QL2+3) group

SUMMARY:
included patients were divided into 4 groups and each group received a mode of post cesarian section analgesia and pain was assessed by visual analogue scale at rest and movement.

1. st group epidural analgesia
2. nd group Quadratus lumborum type 2
3. rd group Quadratus lumborum type 3
4. th group Quadratus lumborum type (2+3)

DETAILED DESCRIPTION:
Patients fulfilling the eligibility criteria were approached prior to delivery. The attending physician explained the nature of the study and all patients signed an informed consent then patients were divided in to four groups as follows (equal sample size in each group): the QLB type 2 (QL2 group), QLB type 3 (QL3 group), QLB type 2 +3 (QL2+3 group) and EA only group.

A 16-gauge intravenous cannula pathway was established in the non-dominant hand or arm in the operation unit. All parturient with standard monitoring including electrocardiogram, pulse arterial oxygen saturation, respiratory rate and non-invasive blood pressure (NIBP) was performed combined with spinal and epidural anesthesia before C-section in the left lateral position and peripheral nerve block at the end of surgery by an experienced doctor (A.M.A). The epidural needle was inserted into the lumbar epidural space at the level of L2-3 intervertebral space.

After finding the epidural space using loss of resistance to saline technique, the tip of a spinal needle passed through the epidural needle. To achieve a sensory block height to the level of the sixth thoracic dermatome, every parturient received intrathecal anesthesia of 0.75% bupivacaine (1.3-1.7 )mL. Then, the needle was withdrawn and then an epidural catheter was inserted through the epidural needle in case the failure of intrathecal anesthesia. All surgical treatments were performed successfully in the usual manner.

Immediately after surgery, all subjects were transferred to the post-anesthesia care unit (PACU) and administered pre-determined analgesia, All parturient were lift in the supine position, tilting 45 degrees to the opposed side in order to place the low-frequency convex probe properly and see the sonography clearly. Bilateral QLB was performed using the atraumatic needle (22-G, 120-mm needle for peripheral nerve blocks) advanced in-plane under the guidance of an ultrasound machine. The ultrasonogram of the abdominal wall was displayed clearly through probe moving or tilting. Pillows helped to relieve the tension along the abdominal wall of parturient. The whole procedure was performed strictly according to clinical protocol.

In this study, QL2 or QL3 were conducted through an anterolateral approach with the supine position as mentioned in (Sato et al, 2017). The ultrasound transducer was placed transversely on both flanks at the horizontal level of L2-3 and adjusted until the "Shamrock sign" formed of QL muscle, psoas major and erector spinae was visualized, with imaging depth set between 0 and 9.9 cm. Needles will be penetrated in an anterolateral to posteromedial direction. Local anesthetic will be injected posterior to QL muscle in QL2, while in QL3, it will be located between QL muscle and psoas major. QL2+3 block was conducted in the same plane with only one puncture on each side.

QL2 and QL3 groups received 0.2% ropivacaine at 30 mL at the sites mentioned above in each side for a total of 60 mL. For QL2+3 group, they recieved 0.2% ropivacaine 15 mL at each point of injection with the needle inserting only once in each side. The solution was injected after negative aspiration to exclude vascular puncture. As for the EA group, we used a single bolus of 6 mL saline solution containing 9 mg ropivacaine (0.15%) and 2 mg morphine via the epidural catheter as postoperative analgesia, and meanwhile, they received a procedure like QL2, but only saline was injected as placebo.

Epidural catheters were detached from all parturient after the procedure mentioned above. Parturient received a standard postoperative analgesic regime of regular oral paracetamol 1.0 g 6 hourly.

ELIGIBILITY:
Inclusion Criteria:

* a normal singleton pregnancy lasting at least 37 weeks, body weight (50-70) kg, as well as having an American Society of Anesthesiologists (ASA) physical status I or II

Exclusion Criteria:

* Individuals with a history of congenital coagulopathy, certain infections, or cognitive impairments that would prevent them from using the verbal rating pain score method or the patient-controlled analgesia (PCA) pump were not involved in the study

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The current study is a prospective cohort study that was conducted on (80) patients in Sohag university hospital who were fulfilling the eligibility criteria and presented to the department of Obstetrics and Gynecology at Sohag University hospital (Egyptian tertiary referral hospital) who are requesting immediate postpartum analgesia. The attending physician had explained the nature of the study and all patients included signed an informed consent.
  All participants were subjected to thorough history taking including age, obstetric history, menstrual history, residency, occupation, medical history, surgical history and family history. Clinical examination and full investigations were done as preparation for elective cesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | zero, four, six, twelve, twenty-four hours & forty-eight hours postoperatively
  Total morphine consumption at specified intervals following operation in addition to postoperative pain assessment by the visual analogue scale (VAS, 0-100 mm) at rest and movement

SECONDARY OUTCOMES:
The side effects of the different interventions | four, six, twelve, twenty-four hours & forty-eight hours postoperatively
  Nausea & vomiting as well as itching, weak legs, urine retention, infection & bleeding

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Sohag University, Medical school, Sohag
  - Sohag University hospital, Sohag

IPD SHARING:
Plan to Share IPD: Undecided
Data is available with authors and can be only shared after reasonable request and approval for Sohag medical research committee